CLINICAL TRIAL: NCT05769166
Title: Prevalence Of Deleterious Oral Habits Among a Group of School Children in Cairo, Egypt: Cross-Sectional Study
Acronym: ACU333
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf A.Elsabour, Teaching assistant, Ahram Canadian University
Other Study IDs: ACU 333
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Habits; Bruxism; Sucking Behavior; Nail Biting
MeSH Terms: conditions — Habits; Bruxism; Sucking Behavior; Nail Biting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School children: school children aged from five to seven years
  Interventions: Other: thired domain of nordic orofcial test-screen

INTERVENTIONS:
Other: thired domain of nordic orofcial test-screen — its a questionnaire which the parent will answer

SUMMARY:
This study aims to detect the prevalence of practicing oral habits among a group of school children in Cairo, Egypt.

DETAILED DESCRIPTION:
An online questionnaire utilizing the third domain of Nordic Orofacial Test screen will be distributed among school children (aged five to seven years) parents to measure the prevalence of oral habits.

ELIGIBILITY:
Inclusion Criteria:

* school children
* accept to participate
* children within the age group

Exclusion Criteria:

* special health care needs children

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school children aged from five to seven years
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
oral habits (presence / absence) | baseline record
  practicing one or more of the following habit(s): sucking habits, nail biting, bruxism